CLINICAL TRIAL: NCT06022848
Title: Does Occipital Nerve Stimulation Alter Pain Response as Measured by Quantitative Sensory Testing in Patients With Chronic Migraine or Cluster Headache
Brief Title: Quantitative Sensory Testing and Occipital Nerve Stimulator
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 210723
Record Dates: First submitted 2019-06-28; First posted 2023-09-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Migraines
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quantitative sensory testing (Experimental)
  Interventions: Procedure: occipital nerve stimulator

INTERVENTIONS:
Procedure: occipital nerve stimulator — Quantitative sensory testing
  Other Names: Quantitative sensory testing

SUMMARY:
The primary aim of this study is to assess the reversibility of a range of psychophysical markers of pain processing in patients with chronic migraine or cluster headache before and after ONS insertion and comparing to patients having a general anaesthetic (GA) for a non-painful aetiology at Barts Health NHS Trust. We will also compare with healthy volunteers not undergoing surgery.

To establish whether pain perception alters in patients with chronic migraine/cluster headache having ONS using questionnaires and compare to patients having a general anaesthetic for a non- painful procedure D & C at Barts Health NHS Trust.

Are pain markers (Glutamate, TGF-B1) altered with ONS?

DETAILED DESCRIPTION:
Headache is one of the most common neurological problems accounting for 4% of primary care consultations and up to 30% of neurology appointments. Even though considerable advances in the understanding of the pathogenesis of migraine, new pharmacologic treatments and the emergence of new innovative interventions for difficult cases, in many patients with migraine remain intractable to medical therapy.

The trigeminocervical complex (TCC) has a crucial role in the pathophysiology of migraines. The TCC is a common convergent pathway by which both trigeminal (dural) and cervical (mainly via the greater occipital nerve) afferent inputs project into higher centres in the thalamus and cortex. This afferent pathway is further influenced by the conditioned pain modulation (CPM) pathway originating from the brainstem structures including periaqueductal grey matter, nucleus raphe magnus, and the rostroventral medulla. There is some evidence to suggest that increased peripheral sensitization of the afferent inputs of the TCC, generalized central sensitization of the trigemino-spinal or the second order trigeminal neurons and impaired descending pain inhibitory pathway, may all contribute to the development of the chronic intractable or treatment resistant primary headache disorder Neurostimulation techniques for treating intractable headache range from invasive deep brain stimulation to less invasive peripheral implantation and stimulation. In 1999 Weiner and Reed described the beneficial effects of subcutaneous Occipital nerve stimulation (ONS) in patients with medically intractable, highly disabling chronic headache disorders Open-label studies have suggested that this treatment modality is effective and safe (Lambru and Matharu 2012). Although the exact mechanism of action is poorly understood, ONS is thought to act by stimulating the distal branches of C1, C2 and C3 in turn influencing the TCC favourably by inhibiting the nociceptive process, resulting in an improvement of symptoms. Previous work has demonstrated a consistent and sustained improvement in conditioned pain modulation (CPM) following ONS as confirmed with quantitative sensory testing (QST) (Wodehouse et al, 2014). QST has the particular advantage of being a functional test that provides a quantitative pain stimulus and assesses the subject's individual response to the stimulus. QST also provides a reliable assessment of changes in pain thresholds and the benefit of ONS. However general anaesthetic has also been demonstrated to cause changes/improvements in pain thresholds, peripheral and central sensitisation and this effect can be long lasting and may account for changes/improvements as measured by QST in subjects having ONS that the anaesthetic provides relief as opposed to the ONS intervention.

Quantitative sensory testing (QST) QST is a term used to describe different forms of psychophysical testing of skin, mucosa, or muscle tissue that assess sensory and pain perception pathways. Nociception inputs can trigger a prolonged but reversible increase in the excitability and synaptic efficacy of neurons in central nociceptive pathways, the phenomenon of central sensitisation in turn manifesting as pain hypersensitivity, particularly dynamic tactile allodynia, and secondary punctate or pressure hyperalgesia and enhanced temporal summation.

QST has been used for measuring thresholds for different sensations in neuropathic pain reflecting the possible nerve fibres that may be implicated in the pathogenesis. Heat sensation threshold reflects the unmyelinated C-fiber function, cold sensation threshold reflects the thinly myelinated A-fiber function and vibration threshold reflects the thickly myelinated AB- fiber function.

QST tests can be classified into the following:

Measurement of pressure pain thresholds (PPT) (Static measure): This test measures sensitivity of peripheral pain pathways to increasing mechanical pressure. A computer-controlled pressure algometer (available as a bed side instrument) is used to measure PPTs at a standardized point and compared with the affected area. A standardized speed of pressure increase of 0.3kg/s is kept constant during pressure application to the point when perception changes from pressure to pain (pressure pain threshold). This is useful for confirming small fibres neuropathic lesion.

Temperature thresholds: Thermal QST evaluates small nerve fibres, using thresholds for warm, cold, heat-induced pain and cold-induced pain. It involves altering a thermal stimulus until a sensation is perceived. Four sensory sub-modalities will be measured; C fibre mediated warm sensation (WS), A-delta fibre mediated cold sensation (CS), heat induced pain (HP) (mostly C fibre mediated sensation with some involvement of A-delta fibres) and C- and A-delta fibre mediated cold induced pain (CP).

Measurement of central sensitisation (Dynamic measure):

This will be done using 2 different techniques as outlined below.

1. Conditional Pain Modulation: Activity within the spinal dorsal horn arising from peripheral nociceptive inputs can be modulated by powerful descending inhibitory and facilitatory mechanisms. An example is provided by the phenomenon of conditioned pain modulation (CPM), also known as diffuse noxious inhibitory control (DNIC) or heterotrophic noxious conditioning stimulation. This refers to an altered response to a painful stimulus following the administration of a second conditioning stimulus.

   CPM provides one of the main supraspinal pain inhibitory pathways and are impaired in neuropathic pain. Diffuse noxious inhibitory controls refers to the observation that the activity of multi-receptive neurons of the spinal cord can be strongly suppressed by an intensive pain stimulus outside their peripheral receptive field. Induction of CPM can be done by immersion in ice water (so-called cold-pressor test), or hot water on a different/distant body part than the one on which the pain perception testing is being performed. This effect represents a well-established model of endogenous pain modulation.
2. Measurement of Temporal summation- Repetitive delivery of a painful stimulus leads to an increased perception of pain which can be used as a marker for central sensitization. Seventeen, progressively rigid, monofilament, von Frey fibers (filaments represent stimuli from 0.039 - 4386mN) will be used on a standardised position on the back decided by the physician. A baseline NRS score will be obtained from the patient. The von Frey Fibre will first ascertain the least force that measures a sensation of touch or pain (pressure pain threshold). The exact threshold is found by repetitive testing using the ascending fibre sizes. The repetitive stimulation consists of 10 repetitions of a pressure stimulus applied for 1 second duration for 60 seconds. The magnitude of the stimulus is set at the level of the subjects' pressure pain threshold. Patients rate the pain intensity on a NRS for each pressure stimulus, and then for 15 sec after cessation of 10 stimulations.

Clinical Data for QST QST measurements have been used world-wide in the assessment of altered pain experience and have been demonstrated to be safe and well tolerated. There exists published evidence of QST measurements in chronic pain conditions like osteoarthritis, fibromyalgia, migraine and other neuropathic pain conditions.

QST measurements have been used worldwide in the assessment of altered pain experience and have been demonstrated to be safe and well tolerated. We do not expect any risks associated with the QST. Any discomfort experienced is transient and patients at all times are in control with the experience and can stop at any-time.

In addition, there is evidence to suggest that cytokines induce headache and headache pain. Furthermore a higher level of cytokines can stimulate the activation of trigeminal nerves, trigeminal nerve fibre sensitisation, the release vasoactive peptides or other biochemical mediators like nitric oxide, which results in inflammation. Many studies have investigated the role of different cytokines in the pathogenesis of migraine but the results remain controversial. One reason for this may be the differing times of measured cytokines in some cases ictally in others interictally. For this study we propose to takes samples at baseline and at the follow up visits and investigate whether there is any alteration in levels of cytokines with the ONS. We will be focusing on transforming growth factor-beta 1 (TGF-1), which is a multifunctional proinflammatory cytokine involved in the modulation of cell growth, differentiation and repairs following injury and immune modulation. Ishizaki et al., 2005 demonstrated that serum levels of TGF-1 were higher in migraine than in controls. TGF-1 has been described as a platelet-derived cytokine as human platelets contain quantities of dormant TGF-1 and reports have suggested that platelets play an important role in migraine and therefore maybe in involved in headache pathogenesis and development of migraines.

Glutamate is a prominent neurotransmitter and has been implicated in migraine pathogenesis. Migraine pain-relay centers, including the trigeminal ganglion, trigeminal nucleus caudalis, and thalamus, contain glutamate-positive neurons, and glutamate activates the trigeminal nucleus caudalis. Glutamate is implicated in cortical spreading depression, trigeminovascular activation, and central sensitization. Glutamate in blood (plasma) and urine will be measured prior to and after ONS.

ELIGIBILITY:
Inclusion criteria

Subject satisfies standard criteria in the study centre for ONS implantation and the NICE 452 criteria for intractable chronic migraine or cluster headache.

Patients who have given their written informed consent.

Patient is able and willing to comply with study procedures and follow up schedule.

Participants will need a good understanding of the English Language and hence. This is a requirement not just for this research but also for the success of the interventions and the full understanding of QST.

Patients undergoing surgery (non-painful complaint) 'dilatation and curettage' (D&C).

Exclusion criteria

* Any inclusion criteria not met
* Female patients of childbearing age who is or plans on becoming pregnant during the course of the study
* Patients with diabetes
* Patients known to have a condition that in the investigator's judgment precludes participation in the study.
* Patients who have received an investigational drug or have used an investigational device in the 30 days preceding to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reversibility of a range of psychological markers of pain processing in patients with chronic migraine/cluster headache before and after ONS. | 4 WEEKS
  Change QST

SECONDARY OUTCOMES:
Percentage of participants with pain markers (glutamate, TGF-B1) altered with ONS | 12 months
  PAIN MARKERS ALTERED
Number of participants whose functionality and quality of life following ONS - HIT6, | 4 weeks and 12 months
  Q of L change with ONS
The effect on functionality and quality of life following ONS - SF-12v2. | 4 weeks and 12 months
  Q of L change with ONS
The effect on functionality and quality of life following ONS - HAD | 4 weeks and 12 months
  Q of L change with ONS

CONTACTS AND LOCATIONS:
Overall Officials: Vivek mehta, FRCA MD, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No